CLINICAL TRIAL: NCT01886287
Title: Phase II Study of Above-Label Octreotide-LAR in Patients With Insufficiently Controlled Carcinoid Syndrome
Brief Title: P:II Above-Label Octreotide-LAR With Insufficiently Controlled Carcinoid Syndrome
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Slow accrual
Sponsor: H. Lee Moffitt Cancer Center and Research Institute (Other)
Collaborators: Novartis (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: MCC-17410; CSMS995AUS64T (Other: Novartis)
Record Dates: First submitted 2013-06-21; First posted 2013-06-25 (Estimated); Results first posted 2015-01-12 (Estimated); Last update posted 2015-01-12 (Estimated); Status verified 2015-01

CONDITIONS: Neuroendocrine Carcinoma
Keywords: endocrine system; neuroendocrine tumors; neuroendocrine cancer; metastatic; neuroendocrine; gastrointestinal (GI); high-dose octreotide; flushing; diarrhea; quality of life in patients; disease-related symptoms
MeSH Terms: conditions — Carcinoma, Neuroendocrine; Neuroendocrine Tumors; Neoplasm Metastasis; Flushing; Diarrhea

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Octreotide Long-acting Release (LAR) (Experimental): Octreotide LAR will be administered at a dose of 60 mg intramuscularly (IM) every 4 weeks.
  Interventions: Drug: Octreotide LAR

INTERVENTIONS:
Drug: Octreotide LAR — Octreotide LAR as outlined in Treatment Arm.
  Other Names: Sandostatin LAR®

SUMMARY:
The primary purpose of the study is to investigate the effects of high-dose octreotide on flushing, diarrhea, and quality of life in patients whose disease-related symptoms are inadequately controlled by the maximum approved dose of octreotide LAR.

DETAILED DESCRIPTION:
The study population will consist of patients with advanced (metastatic or unresectable) neuroendocrine tumors with suboptimally controlled carcinoid syndrome. While the majority of patients will have primary tumors of the ileocecum (midgut), any serotonin-producing neuroendocrine tumors will be eligible (including pancreatic, lung and unknown primary).

All patients will be followed for adverse events and serious adverse events for 28 days following the last dose of above-label octreotide, or until resolution or stabilization of the event, whichever comes first.

ELIGIBILITY:
Inclusion Criteria:

* Metastatic neuroendocrine tumors that are considered well or moderately differentiated (or low to intermediate grade). Patients with poorly differentiated neuroendocrine carcinomas or small cell carcinomas are excluded from the study.
* Elevated urine 5-hydroxyindoleacetic acid (5-HIAA)
* More than 2 bowel-movements per day OR more than 4 flushing episodes per week on average
* Patient currently on octreotide LAR 30mg every 3 or 4 weeks (for at least 3 cycles prior to screening)
* Age ≥ 18 years
* Minimum of four weeks since any major surgery, liver-directed therapy (embolization, etc.) or systemic cancer treatment other than octreotide LAR
* Eastern Cooperative Oncology Group (ECOG) performance status ≤2
* Life expectancy > 12 weeks
* Reliable contraception should be maintained throughout the study and for 3 months after study drug discontinuation.
* Signed informed consent to participate in the study must be obtained from patients after they have been fully informed of the nature and potential risks by the investigator (or his/her designee) with the aid of written information.

Exclusion Criteria:

* Known hypersensitivity to somatostatin analogues
* Patients with poorly differentiated neuroendocrine cancers
* Patients with liver cirrhosis
* Patients receiving hemodialysis or peritoneal dialysis
* Patients with cachexia who, in the opinion of the investigator, may have difficulty tolerating intramuscular injection
* Patients with symptomatic cholelithiasis or biliary events within past five years (who have not undergone cholecystectomy)
* Patients with recent history (within 5 years) of pancreatitis
* Patients with uncontrolled diabetes (HgA1c >8.0 despite adequate therapy)
* Women of child-bearing potential, UNLESS they are using two birth control methods
* Women who are pregnant or lactating
* HIV positive patients
* History of sustained ventricular tachycardia, ventricular fibrillation, advanced heart block, idiopathic syncope thought to be related to ventricular arrhythmia, or congenital long QT syndrome
* Risk factors for Torsades de Pointes such as cardiac failure, clinically significant/symptomatic bradycardia
* Patients who have any severe and/or uncontrolled medical conditions or other conditions that could affect their participation in the study
* History of noncompliance to medical regimens or unwillingness to comply with the protocol
* Patients who were unable to tolerate or did not benefit from above-label dose octreotide (>30mg) in the past
* Concomitant use of other cancer treatments or carcinoid syndrome treatments (whether standard or experimental). Patients should discontinue any concomitant cancer medications more than two weeks prior to screening.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 2 (Actual)
Dates: Start 2013-12; Primary Completion 2014-08 (Actual); Study Completion 2014-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jonathan Strosberg, M.D., Principal Investigator — H. Lee Moffitt Cancer Center and Research Institute
Locations (1):
- H. Lee Moffitt Cancer Center and Research Institute, Tampa, Florida, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This study was open to accrual at Moffitt Cancer Center 12/10/2013 through 10/10/2014.
Period: Overall Study
Arm/Group | Octreotide Long-acting Release (LAR)
Started | 2
Completed | 0
Not Completed | 2
Not completed — Radiographic disease progression | 1
Not completed — Clinical progression due to disease | 1

BASELINE CHARACTERISTICS:
Population: All participants
Arm/Group | Octreotide Long-acting Release (LAR)
Number analyzed (Participants) | 2
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 1
  >=65 years | 1
Age, Continuous [Median (Full Range); unit: years] | 63 [53 to 73]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0
  Male | 2
Region of Enrollment [Number; unit: participants]
  United States | 2

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Improved Frequency of Diarrhea
Description: The frequencies of flushing, diarrhea, and carcinoid syndrome control rating (scale 1-5) will be measured and compared at week 0 and week 12 . These measurements will be compared using two-sided non-parametric paired Wilcoxon signed-rank.
Time Frame: At 12 weeks
Population: Participants on study at 12 weeks
Measure: Number; unit: participants
Arm/Group | Octreotide Long-acting Release (LAR)
Number analyzed (Participants) | 1
participants | 1

2. Secondary Outcome: Rate of Progression Free Survival (PFS) at 6 Months
Description: Progression-free survival, defined as rate of patients alive and free of progression from the date of first study treatment to the end of trial at 6 months. Progressive disease (PD): at least a 20% increase in the sum of the longest diameter of target lesions, taking as reference the smallest sum longest diameter recorded since the treatment started or the appearance of one or more new lesions.
Time Frame: At 6 months
Population: Evaluable participants on study at 6 months
Arm/Group | Octreotide Long-acting Release (LAR)
Number analyzed (Participants) | 0

ADVERSE EVENTS:
Time Frame: 3 months
Arm/Group | Octreotide Long-acting Release (LAR)
Serious Adverse Events (participants affected / at risk) | 0/2
Other Adverse Events (participants affected / at risk) | 2/2
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Octreotide Long-acting Release (LAR) (N=2)
Edema limbs (General disorders) | 1 (1) — unrelated
Edema trunk (General disorders) | 1 (1) — unrelated
Fatigue (General disorders) | 1 (1) — unrelated
Blood bilirubin increased (Investigations) | 1 (1) — unrelated
Weight loss (Investigations) | 1 (1) — unrelated
Hyperglycemia (Metabolism and nutrition disorders) | 1 (1) — possibly related
Hyperkalemia (Metabolism and nutrition disorders) | 1 (1) — unrelated
Hypokalemia (Metabolism and nutrition disorders) | 1 (1) — unrelated
Anemia (Blood and lymphatic system disorders) | 1 (1) — unrelated
Nausea (Gastrointestinal disorders) | 1 (1) — unrelated
Vomiting (Gastrointestinal disorders) | 1 (1) — unrelated
Bruising (Injury, poisoning and procedural complications) | 1 (1) — unrelated
Hypertension (Vascular disorders) | 1 (1) — unrelated

LIMITATIONS AND CAVEATS:
This study was closed early due to slow accrual. There were no evaluable participants at 6 months for the planned Progression Free Survival measure.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes